CLINICAL TRIAL: NCT06234410
Title: Cardiovascular Risk Assessment For Kidney Transplantation - Utility of Computed Tomography Coronary Angiography in the Assessment of Patients Awaiting Kidney Transplantation
Acronym: CRAFT-CTCA
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); University of Glasgow (Other); NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: TCS/22/09
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Kidney Transplant; Complications
Keywords: Coronary artery disease; Kidney transplantation; Cardiovascular risk assessment; Heart disease; Chronic kidney disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma (including for potential genetic analysis) will be taken from participants and stored.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients waitlisted for kidney transplantation: Patients who have been placed on the waiting list for a kidney transplant within Scotland
  Interventions: Radiation: Computed tomography coronary angiography (CTCA)

INTERVENTIONS:
Radiation: Computed tomography coronary angiography (CTCA) — Single CTCA scan prior to kidney transplantation

SUMMARY:
Cardiovascular disease (for example, heart attack, stroke, heart failure) is the commonest complication of kidney failure. Kidney transplantation reduces cardiovascular risk but cardiovascular disease remains the commonest cause of death in patients following transplantation.

Current strategies to assess patient's cardiovascular risk prior to kidney transplantation do not identify those at highest risk and do not improve outcomes.

This study will use a heart scan known as computed tomography coronary angiography (CTCA) to see whether this scan can identify patients at highest risk of future cardiovascular disease prior to transplantation. Studies have shown it is able to do this in patients with normal kidney function.

The aim of this study is to develop CTCA as an effective tool to risk stratify patients prior to kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Has kidney failure and is on the waitlist for a kidney transplant
* Age 16 years and over
* Able to give informed consent

Exclusion Criteria:

* Contraindication to CT scanning, including contrast allergy
* Patients being considered for a simultaneous kidney-pancreas, kidney-liver and/or kidney-islet transplantation
* Inability to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on the kidney transplant waitlist
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have either a myocardial infarction or cardiovascular death | From time of CTCA scan to 36- and 60-months follow-up
  The first event of myocardial infarction or cardiovascular death

SECONDARY OUTCOMES:
Number of participants who have a fatal or non-fatal myocardial infarction | From time of CTCA scan to 36- and 60-months follow-up
  The first event of myocardial infarction (MI). MI will be defined according to the 4th Universal Definition of Myocardial Infarction.
Number of participants who are hospitalised due to any cardiovascular event | From time of CTCA scan to 36- and 60-months follow-up
  Hospital admission due to any cardiovascular event (including myocardial infarction, heart failure, stroke, or any other cardiovascular disease)
Number of participants who die (all-cause death) | From time of CTCA scan to 36- and 60-months follow-up
  Death due to any cause
Number of participants who have a cardiovascular death | From time of CTCA scan to 36- and 60-months follow-up
  Death due to a cardiovascular cause (including myocardial infarction, heart failure, stroke, or any other cardiovascular disease)

OTHER OUTCOMES:
Number of participants who suffer a clinically significant acute kidney injury following study CTCA scan | From time of CTCA scan to 28 days follow-up
  Unexpected progression to dialysis (haemodialysis or peritoneal dialysis) within 28 days of study CTCA scan
Number of participants who have clinically significant abnormal non-cardiac findings on study CTCA scan | From time of CTCA scan to 12 months follow-up
  Abnormal non-cardiac findings (e.g., lung mass), not related to a pre-existing condition and requiring further investigation

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MBChB, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - Queen Elizabeth Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the primary paper, a deidentified individual participant data set will be will be made available for data sharing purposes, subject to necessary governance approvals. Access to the deidentified dataset will be under a controlled access model.